CLINICAL TRIAL: NCT00782158
Title: Hepatitis B and HIV Co-Infection in Uganda
Brief Title: Hepatitis B and HIV Co-Infection in Patients in Uganda
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909016; 09-I-N016
Record Dates: First submitted 2008-10-29; First posted 2008-10-31 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2018-12-14

CONDITIONS: Hepatitis B; HIV Infections
Keywords: HIV; Hepatitis B; Coinfection; Liver Fibrosis; Transient Elastography
MeSH Terms: conditions — Hepatitis B; HIV Infections; Coinfection; Liver Cirrhosis

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This study will determine the amount of liver scarring (fibrosis) or liver damage in people infected with 1) hepatitis B virus (HBV, a virus that can infect the liver); 2) HIV (the virus that causes AIDS); 3) both HBV and HIV; and 4) neither HBV nor HIV. Liver fibrosis and liver damage can have many causes, including alcohol, certain medicines, exposure to some contaminated foods and infections with viruses that affect the liver (such as HBV). About 25 million people in sub-Saharan Africa are infected with HIV and about 50 million with chronic HBV, yet very little information is available on how many people are infected with both viruses and the medical implications of co-infection.

Participants in Uganda s Rakai Health Sciences Program (RHSP) or Infectious Diseases Institute (IDI) clinic who are 18 years of age or older may be eligible for this study.

People enrolled in the study come to the clinic for at least one visit and may be asked to return yearly. During the visit, participants undergo the following procedures:

* Questionnaire and a short interview about their health and quality of life.
* Physical examination and blood draw. The blood is tested for HBV and other factors that may suggest liver disease. Blood drawn at previous clinic visits or from other studies may also be tested.
* Liver evaluation using a FibroScan, a medical device that uses elastic waves to measure liver stiffness in a process similar to ultrasound scanning. For this test, the subjects lies flat on the back with the arm extended out. The tip of the machine s probe is covered with gel and placed on the skin between the ribs at the level of the right lobe of the liver. The machine produces a little tap on the skin that sends a wave out and checks how fast the wave moves. The speed of the wave indicates the amount of scarring in the liver.

DETAILED DESCRIPTION:
While there are around 25 million HIV-infected persons in sub-Saharan Africa, there are also an estimated 50 million with chronic hepatitis B virus (HBV) infection. Yet data from Africa on the prevalence and clinical implications of HIV/HBV co-infection are sparse or unavailable. The scale-up of' HIV treatment with antiretroviral medication (ARVs) in Africa, should result in substantial reductions in morbidity and mortality. In developed countries, however, improved survival with highly active antiretroviral therapy (HAART) has been associated with notable increases in mortality due to liver disease among HIV-infected persons. Also, persons co-infected with hepatitis viruses have significantly higher liver-related toxicity with ARVs compared to persons infected with HIV alone. Our protocol will investigate predictors of liver disease among co-infected participants. The proposed study directly addresses the problem of HIV/HBV co-infection by examining the association of HBV viral markers with the development of significant liver fibrosis (defined by transient elastography). In addition to strengthening the clinical research capacity of our Ugandan colleagues, completion of our study aims will provide needed information for understanding the complex interaction of HBV and HIV, for projecting the future burden of liver disease related to the HIV epidemic, for clinical management of HBV infection in the setting of co-infection with HIV, and for optimizing the benefits while mitigating the potential deleterious consequences of antiretroviral programs in Africa.

Serological screening will be performed on up to 11,000 subjects in order to identify up to 2,400 subjects to be recruited into the clinical protocol. All people who choose to participate in the study will be asked to come to the clinic for at least 1 visit. If continuing funding is obtained, participants may be asked to return for additional yearly follow-up visits.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Willing and able to provide individual informed consent
  2. Currently being followed at the RHSP or IDI Adult Infectious Disease Clinic
  3. Persons aged 18 years and older

EXCLUSION CRITERIA:

1. Age less than 18 years
2. Women who are pregnant
3. Participants with a cardiac device (i.e., pacemaker)
4. Participants not willing to allow storage of samples
5. Participants not able to follow study instructions

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6303 (Actual)
Dates: Start 2008-10-27; Study Completion 2018-12-14

PRIMARY OUTCOMES:
Liver fibrosis and hepatoxicity

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Reynolds, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- Uganda (2):
  - Infectious Diseases Institute, Kampala
  - International Ctr for Excellence in Research and Rakai Health Sciences Program, Rakai

REFERENCES:
- [Background] Stabinski L, Reynolds SJ, Ocama P, Laeyendecker O, Ndyanabo A, Kiggundu V, Boaz I, Gray RH, Wawer M, Thio C, Thomas DL, Quinn TC, Kirk GD; Rakai Health Sciences Program. High prevalence of liver fibrosis associated with HIV infection: a study in rural Rakai, Uganda. Antivir Ther. 2011;16(3):405-11. doi: 10.3851/IMP1783. PMID 21555823
- [Background] Auerbach BJ, Reynolds SJ, Lamorde M, Merry C, Kukunda-Byobona C, Ocama P, Semeere AS, Ndyanabo A, Boaz I, Kiggundu V, Nalugoda F, Gray RH, Wawer MJ, Thomas DL, Kirk GD, Quinn TC, Stabinski L; Rakai Health Sciences Program. Traditional herbal medicine use associated with liver fibrosis in rural Rakai, Uganda. PLoS One. 2012;7(11):e41737. doi: 10.1371/journal.pone.0041737. Epub 2012 Nov 27. PMID 23209545
- [Background] Redd AD, Wendel SK, Grabowski MK, Ocama P, Kiggundu V, Bbosa F, Boaz I, Balagopal A, Reynolds SJ, Gray RH, Serwadda D, Kirk GD, Quinn TC, Stabinski L. Liver stiffness is associated with monocyte activation in HIV-infected Ugandans without viral hepatitis. AIDS Res Hum Retroviruses. 2013 Jul;29(7):1026-30. doi: 10.1089/aid.2013.0004. Epub 2013 May 8. PMID 23548102